CLINICAL TRIAL: NCT02340897
Title: Diagnostic Accuracy and Inter-rater Agreement of Chest Computed Tomography in the Diagnosis of Nontuberculous Mycobacterial Lung Disease
Brief Title: Diagnostic Accuracy of Nontuberculous Mycobacterial Lung Disease Based on Chest CT
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Joon Yim, Professor, Seoul National University Hospital
Other Study IDs: 2014-1043
Record Dates: First submitted 2014-12-27; First posted 2015-01-19 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Mycobacterium Infections, Nontuberculous
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Nontuberculous lung disease: Patients with Nontuberculous Mycobacteria satisfying American Thoracic Society and British Thoracic Society guidelines
- pulmonary tuberculosis: Patients with culture confirmed tuberculosis
- bronchiectasis: Patients with bronchiectasis based on chest CT findings as well as symptoms

SUMMARY:
The aim of this study was to elucidate the accuracy and inter-rater agreement of diagnosis of nontuberculous mycobacterial lung disease based on chest computed tomography findings.

DETAILED DESCRIPTION:
To elucidate the accuracy and inter-rater agreement of diagnosis of nontuberculous mycobacterial lung disease based on chest CT, two pulmonologists and two chest radiologists were requested to interpret chest CT of patients nontuberculous mycobacterial lung disease satisfying diagnostic criteria of American Thoracic Society as well as British Thoracic Society, or pulmonary tuberculosis. Two pulmonologists and two chest radiologists > 10 years of clinical experiences at a tertiary referral hospital participated as raters in this study. They were blinded to the any clinical information of the patients including the specific diagnosis, except age and sex. The interpretations of four raters were analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Nontuberculous mycobacterial patients satisfying diagnostic criteria suggested by American Thoracic Society
* Patients with bacteriologically confirmed pulmonary tuberculosis
* Patients with bronchiectasis, confirmed by clinically as well as radiographically

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with nontuberculous mycobacterial lung diseases, pulmonary tuberculosis, bronchiectasis
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity for the diagnosis of nontuberculous mycobacterial lung disease | baseline
  Percentage of cases diagnosed as nontuberculous mycobacterial lung disease by four raters out of confirmed cases with nontuberculous mycobacterial lung disease

SECONDARY OUTCOMES:
Inter-rater correlation (kappa value) for the diagnosis of nontuberculous mycobacterial lung disease | baseline
  Inter-rater correlation between four raters
Specificity for the diagnosis nontuberculous mycobacterial lung disease | baseline
  Percentage of cases diagnosed as other than nontuberculous mycobacterial lung disease by four raters out of confirmed cases with other than nontuberculous mycobacterial lung disease

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, Principal Investigator — Seoul National University Hospital